CLINICAL TRIAL: NCT01191203
Title: Prospective Assessment of Acceptability and Adherence Associated With Use of the Copper Intrauterine Device (CuT380A-IUCD) Compared to Depo-medroxyprogesterone Acetate (DMPA) Among HIV Positive Women in Lilongwe, Malawi
Brief Title: Randomized Control Trial Copper Intrauterine Device and Depo-medroxyprogesterone Acetate (DMPA) of HIV+ Women in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of North Carolina (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Lisa Haddad, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00037535
Record Dates: First submitted 2010-06-02; First posted 2010-08-30 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: HIV
Keywords: Acceptability and Adherence to methods
MeSH Terms: interventions — Intrauterine Devices, Copper; Medroxyprogesterone Acetate; N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depo Medroxyprogesterone Acetate (Active Comparator)
  Interventions: Drug: Depo Medroxyprogesterone acetate
- Copper IUD (CuT360) (Active Comparator)
  Interventions: Drug: Copper IUD

INTERVENTIONS:
Drug: Copper IUD — Copper IUD (CuT360)
  Arms: Copper IUD (CuT360)
Drug: Depo Medroxyprogesterone acetate — DMPA 150 mg IM q 3 months
  Other Names: DMPA; Depo Provera
  Arms: Depo Medroxyprogesterone Acetate

SUMMARY:
The IUD is an extremely effective method of contraception yet few women use it worldwide. Considered safe to use in HIV+ women, few studies have evaluated its use among those using antiretroviral therapy. The only prior randomized trial looking at the IUD compared to hormonal contraception noted a high rate of IUD discontinuations. Understanding IUD acceptability and continuation is critical to improve utilization.

* Objective 1: Determine WHO medical eligibility and the willingness for IUD placement
* Objective 2: Compare method-related side effects and adverse events
* Objective 3: Assess the 1-year acceptability and continuation rates

Methods: To address our objectives the investigators have designed a two Phase Study:

* A cross-sectional screening to evaluate contraceptive medical eligibility and desirability
* A randomized controlled trial that will compare acceptability and adherence to DMPA compared to the Copper IUD: enrolling 200 women stable on antiretroviral therapy to follow for 1 year

ELIGIBILITY:
Inclusion Criteria:

* Can provide informed consent
* Women ages 18-45
* Known HIV + status on antiretroviral therapy for at least 6 months
* Not currently pregnant
* Willing to initiate either DMPA or CuT380A-IUD. Women currently using DMPA or CuT380A-IUD will be excluded
* Do not desire to become pregnant within next 12 months
* Intend to stay in Lilongwe region for the duration of the study
* No known uterine anomalies based upon history
* Greater than or equal to 4 weeks post partum
* No known or suspected genital tract cancer
* No evidence of current pelvic inflammatory disease or cervicitis. Women with cervicitis at the time of examination will be treated with antibiotics and eligibility will be reassessed at a follow-up visit at least 7 days after treatment
* No pelvic inflammatory disease within prior 3 months
* No contraindications to DMPA or the CuT380A-IUD per the WHO medical eligibility criteria or Malawi National Reproductive Health Service Delivery Guidelines, 2007
* Based on clinical assessment, no condition that would preclude start of study intervention

Exclusion Criteria:

* Women ages younger than18 or older than 45
* Known HIV + status on antiretroviral therapy less than 6 months or not on antiretroviral therapy
* Pregnant
* Uterine anomaly
* Less than 4 weeks post partum
* Suspected genital tract cancer

Inclusion Criteria:

•Current STI or PID

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Adherence | 1 year
  Number of clients continuing with method at 1 year

SECONDARY OUTCOMES:
Adverse Events | 1 year
  -Number of clients who experience adverse events such as pelvic inflammatory disease, lower genital tract infection, and infection related complications, such as abdominal pain, and irregular vaginal bleeding, as well as lower tract infection determined by clinical examination.
  Side effects such as abnormal vaginal discharge, abnormal bleeding, IUCD expulsion, and other side effects, as measured by clinical examination and client self-report.
  -Risk of excessive vaginal bleeding or anemia: determined by self report and hemoglobin level

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Haddad, MD, Principal Investigator — Emory University; Sam Phiri, PhD, Principal Investigator — Lighthouse Trust
Locations (1):
- The Lighthouse Trust, Lilongwe, Lilongwe, Malawi